CLINICAL TRIAL: NCT01900561
Title: Optimizing Veteran-Centered Prostate Cancer Survivorship Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IIR 12-116
Record Dates: First submitted 2013-07-02; First posted 2013-07-16 (Estimated); Results first posted 2019-04-08 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; survivorship; intervention; telemedicine
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IVR Intervention (Experimental): The intervention will consist of two components, both with content design based on established theories for self-management support: 1) automated telephone monitoring of PC survivor symptoms and goals for symptom reduction, based on a patient empowerment approach, and 2) personally tailored newsletters that incorporate elements of CBT to improve survivors' identification with the material, confidence/self-efficacy in symptom management, and to reduce common cognitive distortions related to successful implementation of behavior change. Intervention-group participants will receive four automated assessment and self-management support calls over a 3-month period (at baseline, 1-month, 2-month, 3-months). Information collected during automated phone assessments will be used to construct tailored newsletters, which will be sent following each automated call.
  Interventions: Behavioral: Interactive Voice Response Symptom Management; Behavioral: Tailored Newsletters
- Enhanced Usual Care (No Intervention): Because of the strong evidence documenting symptom burden in PC survivors, the investigators believe that providing control subjects with some information about symptom self-management is warranted. The investigators further believe, based on the investigators' prior experience conducting RCTs, that offering some type of educational material for Veterans randomized to the control arm will increase their willingness to enroll in the study (as opposed to a pure usual care arm where they would not receive any such materials). Therefore, survivors randomized to the control condition will receive written material at the time of enrollment designed to educate them about PC symptoms and symptom management. Material will be approximately six pages in length, also written at or below an 8th grade reading level, and will include a summary of common symptoms experienced by prostate cancer survivors.

INTERVENTIONS:
Behavioral: Interactive Voice Response Symptom Management — The Interactive Voice Response (IVR) system will provide automated telephone monitoring of PC survivor symptoms and goals for symptom reduction, based on a patient empowerment approach.
  Arms: IVR Intervention
Behavioral: Tailored Newsletters — Personally tailored newsletters will incorporate elements of CBT to improve survivors' identification with the material, confidence/self-efficacy in symptom management, and to reduce common cognitive distortions related to successful implementation of behavior change. Information collected during automated phone assessments will be used to construct tailored newsletters, which will be sent following each automated call.
  Arms: IVR Intervention

SUMMARY:
This study will provide much needed information about how to optimize the quality of care and quality of life of Veterans who are survivors of prostate cancer.

DETAILED DESCRIPTION:
Although there are nearly 150,000 prostate cancer survivors in the VA, there has been little research to understand and improve survivorship care for this large population of Veterans. A substantial proportion of prostate cancer survivors in the general population have significant side effects from treatment (surgery or radiation therapy) that often persist for years, including incontinence, erectile dysfunction, and metabolic syndrome, all of which can contribute to decreased quality of life. The investigators' pilot data suggests that VA prostate cancer survivors experience similar or worse symptom burden to that of the general population of survivors. To address the need to improve patient-centered survivorship care management for Veterans with prostate cancer, the investigators propose a 4 year study with two aims: 1) to conduct a randomized controlled trial to compare a personally tailored automated telephone symptom management intervention for improving symptoms and symptom self-management to usual care. The investigators expect that those in the intervention group will have more confidence in symptom self-management and better symptom self-management and prostate cancer quality of life following the intervention, and that these outcomes will translate to more efficient use of services for these Veterans, and 2) to compare utilization of services among those in the intervention group to those in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Veteran patient at one of the four study sites (Ann Arbor VA, Cleveland VA, Pittsburgh VA, St. Louis VA)
* History of treatment for prostate cancer treated by surgery, radiation or androgen deprivation therapy between 1-10 years prior to identification

Exclusion Criteria:

* No phone number on file
* Not able to converse on the telephone in English
* Treated for metastatic disease or non-prostate cancer
* Dementia or other significant mental impairment

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer is a disease which only affects men.
Enrollment: 556 (Actual)
Dates: Start 2015-04-17 (Actual); Primary Completion 2018-02-07 (Actual); Study Completion 2018-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah T Hawley, PhD MPH BA, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (4):
- United States (4):
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - St. Louis VA Medical Center John Cochran Division, St. Louis, MO, St Louis, Missouri
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Telem DA, Dimick J, Skolarus TA. Dissecting Surgeon Behavior: Leveraging the Theoretical Domains Framework to Facilitate Evidence-based Surgical Practice. Ann Surg. 2018 Mar;267(3):432-434. doi: 10.1097/SLA.0000000000002506. No abstract available. PMID 28902665
- [Background] Skolarus TA, Wittmann D, Hawley ST. Enhancing prostate cancer survivorship care through self-management. Urol Oncol. 2017 Sep;35(9):564-568. doi: 10.1016/j.urolonc.2017.05.008. Epub 2017 Jun 13. PMID 28619632
- [Background] Skolarus TA, Metreger T, Hwang S, Kim HM, Grubb RL 3rd, Gingrich JR, Hawley ST. Optimizing veteran-centered prostate cancer survivorship care: study protocol for a randomized controlled trial. Trials. 2017 Apr 18;18(1):181. doi: 10.1186/s13063-017-1925-4. PMID 28420419
- [Result] Skolarus TA, Metreger T, Wittmann D, Hwang S, Kim HM, Grubb RL 3rd, Gingrich JR, Zhu H, Piette JD, Hawley ST. Self-Management in Long-Term Prostate Cancer Survivors: A Randomized, Controlled Trial. J Clin Oncol. 2019 May 20;37(15):1326-1335. doi: 10.1200/JCO.18.01770. Epub 2019 Mar 29. PMID 30925126

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IVR Intervention | Enhanced Usual Care
Started | 278 | 278
Completed | 261 | 269
Not Completed | 17 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IVR Intervention | Enhanced Usual Care | Total
Number analyzed (Participants) | 278 | 278 | 556
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 74 | 88 | 162
  >=65 years | 204 | 190 | 394
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (5.7) | 66.2 (7.1) | 66.7 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 278 | 278 | 556
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 199 | 186 | 385
  Black | 74 | 83 | 157
  Other | 9 | 15 | 24
  Hispanic | 4 | 5 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 278 | 278 | 556

OUTCOME MEASURES:

1. Primary Outcome: The Expanded Prostate Cancer Index (EPIC) - Urinary Health, Irritative
Description: The EPIC is a 26-item measure that assesses symptom burden in four domains: urinary symptoms, bowel symptoms, sexual symptoms and vitality. Each domain has a subscale related to function and bother which together contribute to disease specific quality of life. Each domain has a range of possible scores from 0 to 100, with lower scores indicating worse symptom burden. Lower EPIC scores for any one domain are associated with lower function in that domain and lower QOL. Thus higher symptom burden, which reflects both function and bother scores, translate into lower EPIC scores.
Time Frame: Baseline
Population: Thirty (5.4%) enrollees did not do EPIC-26.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IVR Intervention | Enhanced Usual Care
Number analyzed (Participants) | 264 | 262
score on a scale | 60.1 (28.2) | 61.4 (28.9)

2. Primary Outcome: The Expanded Prostate Cancer Index (EPIC) - Urinary Health, Obstructive
Description: as for outcome 1
Time Frame: Baseline
Population: Thirty (5.4%) enrollees did not do EPIC-26, and two enrollees did only one or two subscales. EPIC-Urinary Health Obstructive was not done in 31 persons.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IVR Intervention | Enhanced Usual Care
Number analyzed (Participants) | 264 | 261
score on a scale | 72.7 (20.0) | 72.5 (20.1)

3. Primary Outcome: The Expanded Prostate Cancer Index (EPIC) - Bowel Health
Description: as for outcome 1
Time Frame: Baseline
Population: Thirty (5.4%) enrollees did not do EPIC-26, and two enrollees did only one or two subscales. EPIC-Bowel Health was not done in 32 persons.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IVR Intervention | Enhanced Usual Care
Number analyzed (Participants) | 264 | 260
score on a scale | 76.5 (21.7) | 77.6 (22.2)

4. Primary Outcome: The Expanded Prostate Cancer Index (EPIC) - Sexual Health
Description: as for outcome 1
Time Frame: Baseline
Population: Thirty (5.4%) enrollees did not do EPIC-26, and two enrollees did only one or two subscales. EPIC-Sexual Health was not done in 58 persons.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IVR Intervention | Enhanced Usual Care
Number analyzed (Participants) | 253 | 245
score on a scale | 21.6 (25.5) | 21.8 (26.3)

5. Primary Outcome: The Expanded Prostate Cancer Index (EPIC) - General Health
Description: as for outcome 1
Time Frame: Baseline
Population: Thirty (5.4%) enrollees did not do EPIC-26, and two enrollees did only one or two subscales. EPIC-General Health was not done in 32 persons.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IVR Intervention | Enhanced Usual Care
Number analyzed (Participants) | 264 | 260
score on a scale | 71.0 (20.9) | 67.9 (21.5)

6. Primary Outcome: The Expanded Prostate Cancer Index (EPIC) - EPIC-26 Mean
Description: The EPIC is a 26-item measure that assesses symptom burden in four domains: urinary symptoms, bowel symptoms, sexual symptoms and vitality. Each domain has a subscale related to function and bother which together contribute to disease specific quality of life. Each domain has a range of possible scores from 0 to 100, with lower scores indicating worse symptom burden. Lower EPIC scores for any one domain are associated with lower function in that domain and lower QOL. Thus higher symptom burden, which reflects both function and bother scores, translate into lower EPIC scores.
  The EPIC-26 mean is the average of the five EPIC subscales.
Time Frame: Baseline
Population: Average of 5 EPIC-26 subscales based on 524 person data (260 in control and 264 in IVR group): 30 (5.4%) enrollees did not do EPIC-26, and two enrollees did only one or two subscales. EPIC-Urinary Health Irritative was not done in 30 persons, Urinary Health Obstructive in 31, Bowel Health in 32, Sexual Health in 58 and General Health in 32 persons
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IVR Intervention | Enhanced Usual Care
Number analyzed (Participants) | 264 | 260
score on a scale | 60.8 (16.5) | 60.9 (16.7)

7. Primary Outcome: The Expanded Prostate Cancer Index (EPIC) - Urinary Health, Irritative
Description: as for outcome 1
Time Frame: 5 Months
Population: N with non-missing data for the specific measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IVR Intervention | Enhanced Usual Care
Number analyzed (Participants) | 242 | 259
score on a scale | 63.4 (29.5) | 61.8 (28.5)

8. Primary Outcome: The Expanded Prostate Cancer Index (EPIC) - Urinary Health, Obstructive
Description: as for outcome 1
Time Frame: 5 Months
Population: N with non-missing data for the specific measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IVR Intervention | Enhanced Usual Care
Number analyzed (Participants) | 241 | 256
score on a scale | 77.4 (19.7) | 74.5 (20.2)

9. Primary Outcome: The Expanded Prostate Cancer Index (EPIC) - Bowel Health
Description: as for outcome 1
Time Frame: 5 Months
Population: N with non-missing data for the specific measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IVR Intervention | Enhanced Usual Care
Number analyzed (Participants) | 240 | 258
score on a scale | 80.6 (19.0) | 79.8 (21.6)

10. Primary Outcome: The Expanded Prostate Cancer Index (EPIC) - Sexual Health
Description: as for outcome 1
Time Frame: 5 Months
Population: N with non-missing data for the specific measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IVR Intervention | Enhanced Usual Care
Number analyzed (Participants) | 221 | 241
score on a scale | 25.8 (26.5) | 25.1 (28.7)

11. Primary Outcome: The Expanded Prostate Cancer Index (EPIC) - General Health
Description: as for outcome 1
Time Frame: 5 Months
Population: N with non-missing data for the specific measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IVR Intervention | Enhanced Usual Care
Number analyzed (Participants) | 240 | 257
score on a scale | 74.8 (21.3) | 71.2 (21.9)

12. Primary Outcome: The Expanded Prostate Cancer Index (EPIC) - Urinary Health, Irritative
Description: as for outcome 1
Time Frame: 12 Months
Population: N with non-missing data for the specific measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IVR Intervention | Enhanced Usual Care
Number analyzed (Participants) | 220 | 221
score on a scale | 62.8 (29.7) | 63.6 (29.3)

13. Primary Outcome: The Expanded Prostate Cancer Index (EPIC) - Urinary Health, Obstructive
Description: as for outcome 1
Time Frame: 12 Months
Population: N with non-missing data for the specific measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IVR Intervention | Enhanced Usual Care
Number analyzed (Participants) | 221 | 219
score on a scale | 76.3 (19.0) | 75.1 (20.0)

14. Primary Outcome: The Expanded Prostate Cancer Index (EPIC) - Bowel Health
Description: as for outcome 1
Time Frame: 12 Months
Population: N with non-missing data for the specific measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IVR Intervention | Enhanced Usual Care
Number analyzed (Participants) | 221 | 220
score on a scale | 79.2 (20.7) | 81.0 (21.7)

15. Primary Outcome: The Expanded Prostate Cancer Index (EPIC) - Sexual Health
Description: as for outcome 1
Time Frame: 12 Months
Population: N with non-missing data for the specific measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IVR Intervention | Enhanced Usual Care
Number analyzed (Participants) | 211 | 208
score on a scale | 29.3 (29.7) | 26.5 (30.9)

16. Primary Outcome: The Expanded Prostate Cancer Index (EPIC) - General Health
Description: as for outcome 1
Time Frame: 12 Months
Population: N with non-missing data for the specific measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IVR Intervention | Enhanced Usual Care
Number analyzed (Participants) | 218 | 218
score on a scale | 75.8 (18.6) | 73.5 (20.7)

17. Primary Outcome: Confidence in Symptom Self-Management
Description: Confidence in symptom self-management was measured using a 5-item scale developed from our pilot work. Scores range from 5 to 15 with higher scores indicating higher level of confidence.
Time Frame: 5 months
Population: N with non-missing data for the specific measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IVR Intervention | Enhanced Usual Care
Number analyzed (Participants) | 235 | 244
score on a scale | 13.1 (2.1) | 13.1 (2.1)

18. Primary Outcome: Confidence in Symptom Self-Management
Description: as for outcome 17
Time Frame: 12 months
Population: N with non-missing data for the specific measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IVR Intervention | Enhanced Usual Care
Number analyzed (Participants) | 206 | 210
score on a scale | 13.5 (1.9) | 12.9 (2.2)

19. Secondary Outcome: Cancer Control
Description: We assessed perceived cancer control and outlook using five items from a validated measure developed to examine the psychosocial impact of prostate cancer. This measure, the Measuring Patients' Perceptions of the Outcomes of Treatment for Early PC instrument by Clark et al., includes three domains related to confidence that one's cancer is under control, worries about recurrence, and appraisals of one's coping with PC. Cancer control was assessed during the five- and 12-month follow-ups using two cancer control items from the instrument. Scores range from 2 to 10 and higher scores indicate higher confidence that cancer is under control.
Time Frame: 5 months
Population: N with non-missing data for the specific measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IVR Intervention | Enhanced Usual Care
Number analyzed (Participants) | 241 | 257
score on a scale | 9.6 (2.1) | 9.6 (2.2)

20. Secondary Outcome: Cancer Control
Description: as for outcome 19
Time Frame: 12 months
Population: N with non-missing data for the specific measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IVR Intervention | Enhanced Usual Care
Number analyzed (Participants) | 223 | 226
score on a scale | 9.4 (1.7) | 9.4 (1.8)

21. Secondary Outcome: Cancer Outlook
Description: We assessed perceived cancer control and outlook using five items from a validated measure developed to examine the psychosocial impact of prostate cancer. This measure, the Measuring Patients' Perceptions of the Outcomes of Treatment for Early PC instrument by Clark et al., includes three domains related to confidence that one's cancer is under control, worries about recurrence, and appraisals of one's coping with PC. Cancer outlook was assessed during the five- and 12-month follow-ups using three cancer outlook items from the instrument. Scores range from 3 to 15 and higher scores indicate more positive cancer outlook.
Time Frame: 5 months
Population: N with non-missing data for the specific measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IVR Intervention | Enhanced Usual Care
Number analyzed (Participants) | 236 | 253
score on a scale | 7.2 (2.2) | 7.3 (2.3)

22. Secondary Outcome: Cancer Outlook
Description: as for outcome 21
Time Frame: 12 months
Population: N with non-missing data for the specific measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IVR Intervention | Enhanced Usual Care
Number analyzed (Participants) | 226 | 224
score on a scale | 7.1 (2.0) | 6.8 (2.2)

23. Secondary Outcome: Perceived Efficacy in Patient-Physician Interactions (PEPPI) - 5-item Short Form
Description: Self-efficacy in patient-physician interactions was assessed at 5 and 12 months using a five-item short form version of the Perceived Efficacy in Patient-Physician Interactions (PEPPI). The PEPPI was developed to measure older patients' self-efficacy in obtaining medical information and attention to their medical concerns from physicians. Scores range from 0-25 with higher scores indicating higher self-efficacy.
Time Frame: 5 months
Population: N with non-missing data for the specific measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IVR Intervention | Enhanced Usual Care
Number analyzed (Participants) | 241 | 254
score on a scale | 21.8 (3.9) | 21.9 (3.8)

24. Secondary Outcome: Perceived Efficacy in Patient-Physician Interactions (PEPPI) - 5-item Short Form
Description: as for outcome 23
Time Frame: 12 months
Population: N with non-missing data for the specific measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IVR Intervention | Enhanced Usual Care
Number analyzed (Participants) | 223 | 220
score on a scale | 21.5 (4.3) | 21.7 (4.5)

25. Secondary Outcome: Brief Cope - 6 Items
Description: We assessed participants' coping during the five- and 12-month follow-up assessments using six items from the 28-item Brief Cope instrument. This instrument measures emotion-focused, problem-focused, and dysfunctional coping and has been used in cancer survivors. Scores range from 1 to 5 with higher scores indicating better coping skills.
Time Frame: 5 months
Population: N with non-missing data for the specific measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IVR Intervention | Enhanced Usual Care
Number analyzed (Participants) | 227 | 248
score on a scale | 2.8 (0.9) | 2.6 (1.0)

26. Secondary Outcome: Brief Cope - 6 Items
Description: as for outcome 25
Time Frame: 12 months
Population: N with non-missing data for the specific measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IVR Intervention | Enhanced Usual Care
Number analyzed (Participants) | 221 | 203
score on a scale | 2.7 (0.9) | 2.6 (1.0)

27. Secondary Outcome: Veteran Quality of Life Scale (VR-12) - Physical Health, 2 Items
Description: We assessed subjective physical health using 2 items from the VR-12 (SF-12 for veterans), an established measure of overall QOL that includes perceptions of one's health that may be impacted by prostate cancer. The scores range from 1- 3 and higher scores correspond to better health.
Time Frame: 12 months
Population: N with non-missing data for the specific measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IVR Intervention | Enhanced Usual Care
Number analyzed (Participants) | 226 | 228
score on a scale | 2.2 (0.7) | 2.3 (0.7)

28. Secondary Outcome: Veteran Quality of Life Scale (VR-12) - Emotional Health, 3 Items
Description: We assessed subjective emotional health using 3 items from the VR-12 (SF-12 for veterans), an established measure of overall QOL that includes perceptions of one's health that may be impacted by prostate cancer. The scores range from 1- 6 and higher scores correspond to better health.
Time Frame: 12 months
Population: N with non-missing data for the specific measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IVR Intervention | Enhanced Usual Care
Number analyzed (Participants) | 226 | 228
score on a scale | 3.7 (0.6) | 3.6 (0.7)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the start of recruitment on 4/17/15 through the final 12-month assessment on 2/2/18.
Arm/Group | IVR Intervention | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 1/278 | 3/278
Serious Adverse Events (participants affected / at risk) | 3/278 | 1/278
Other Adverse Events (participants affected / at risk) | 0/278 | 0/278
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IVR Intervention (N=278) | Enhanced Usual Care (N=278)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0) — Pt was admitted to hospital for previously scheduled left total hip arthroplasty
Subdural hematoma (Nervous system disorders) | 0 (0) | 1 (1) — Patient was admitted to hospital with a subdural hematoma.
Kidney Failure (Renal and urinary disorders) | 1 (1) | 0 (0) — Patient reported that he had been hospitalized for kidney failure.
Stroke (Vascular disorders) | 1 (1) | 0 (0) — Patient suffered a stroke rendering him unable to speak.

LIMITATIONS AND CAVEATS:
Veterans without telephones or the ability to use automated telephone systems could not enroll.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/61/NCT01900561/Prot_SAP_000.pdf